CLINICAL TRIAL: NCT02986750
Title: Influence of Three Different Formulations of Lachrymal Substitutes on Tear Film Thickness and Other Signs and Symptoms in Patients With Moderate to Severe Dry Eye Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LT2258-PIV-0216
Record Dates: First submitted 2016-12-01; First posted 2016-12-08 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental: Patients with dry eye syndrome 1 (Experimental): 40 Patients with dry eye syndrome
  Interventions: Device: Thealoz Duo Eye Drops
- Experimental: Patients with dry eye syndrome 2 (Active Comparator): 40 Patients with dry eye syndrome
  Interventions: Device: Optive Eye Drops
- Experimental: Patients with dry eye syndrome 3 (Active Comparator): 40 Patients with dry eye syndrome
  Interventions: Device: Systane Ultra Eye Drops

INTERVENTIONS:
Device: Thealoz Duo Eye Drops — Manufacturer: Laboratoires Thea, France
  Arms: Experimental: Patients with dry eye syndrome 1
Device: Optive Eye Drops — Manufacturer: Allergan Pharmaceuticals, Ireland
  Arms: Experimental: Patients with dry eye syndrome 2
Device: Systane Ultra Eye Drops — Manufacturer: Alcon Pharma GmbH
  Arms: Experimental: Patients with dry eye syndrome 3

SUMMARY:
Dry eye syndrome is a highly prevalent ocular disease with an increasing incidence in the elderly population. Topically administered lubricants are the basis for treatment of this disease. However, exact information about influence on tear film thickness and corneal residence time of topical lubricants is still sparse, therefore no ideal treatment regimen has been found.

Recently a new method for assessment of tear film thickness based on ultra-high resolution optical coherence tomography (OCT) has become available. The aim of the present study is to assess the influence on tear film thickness of three different formulations of topical lubricants, in particular Thealoz Duo® Eye Drops, Optive® Eye Drops and Systane Ultra® Eye Drops in patients with moderate to severe dry eye disease. In addition, standard tests for dry eye syndrome, such as the ocular surface disease index (OSDI©), Schirmer I test, corneal fluorescein staining and determination of tear break up time (BUT) will be performed to compare the product effects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged over 18 years
2. Signed and dated written informed consent
3. History of dry eye syndrome for at least 3 months
4. Tear Break Up Time (BUT) ≤ 10 seconds or Schirmer I test ≤ 5 mm and ≥ 2mm
5. OSDI ≥ 22
6. Normal ophthalmic findings except dry eye syndrome, ametropia < 6 Dpt.
7. No administration of topical lubricants 24 hours before the screening examination

Exclusion Criteria:

1. Presence of an ocular pathology judged by the investigator as incompatible with the study.
2. Any other clinical relevant ocular abnormality except DES.
3. History of allergy, known hypersensitivity to one of the components: the study medications or Fluorescein.
4. History of known clinically relevant allergy.
5. Medical or surgical history judged by the investigator to be incompatible with the study participation (hepatic or renal insufficiency; all chronic severe organic disease: metabolic, endocrine, neoplasic, haematological disease; severe psychiatric illness, etc.).
6. History of a recent acute illness with a recovery period within the 2 weeks before the inclusion visit (Day 0).
7. Pregnancy, lactation.
8. Pre-menopausal woman who is not using a reliable birth control method (oral contraceptives or coil) or is not surgically sterilised.
9. Participation in any high-speed or water-sports during the study without ocular protection (goggles or glasses).
10. Subject unable to understand the study instructions or unlikely to comply with the study schedule and treatment.
11. Participation in another clinical study in the 4 weeks before the start of the present study or at the same time as the present study.
12. Subject is a ward of court.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02-13 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Change in tear film thickness as measured with Optical Coherence Tomography (OCT) | 10 weeks; at baseline, 10 minutes, 20 minutes, 40 minutes, 60 minutes, 120 minutes and 240 minutes after instillation of eye drops as well as 4 weeks and 8 weeks after the first instillation
  Tear film thickness as measured with Optical Coherence Tomography (OCT) predose and at defined time points after the first instillation, as well as on each study day

SECONDARY OUTCOMES:
Tear Break Up Time (BUT) | 10 weeks
Subjective evaluation of ocular comfort with questionnaire | 10 weeks
Schirmer I test | 10 weeks
OSDI score | 10 weeks
Corneal fluorescein staining (Oxford grading scale) | 10 weeks
Conjunctival hyperemia score | 10 weeks
Efficacy assessment of eye drops by the patient with questionnaire | 10 weeks
  Efficacy of eye drops will be performed by the patient by choosing one of the following options:
  * Very satisfactory
  * Satisfactory
  * Not very satisfactory
  * Unsatisfactory
Efficacy assessment of eye drops by the investigator with questionnaire | 10 weeks
  Efficacy of eye drops will be performed by the investigator by choosing one of the following options:
  * Very satisfactory
  * Satisfactory
  * Not very satisfactory
  * Unsatisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria